CLINICAL TRIAL: NCT03188640
Title: Health-related Quality of Life, Sexuality and Hormone Status After Bariatric Surgery
Brief Title: Bariatric Surgery, Hormones, and Quality of Life
Acronym: OBLIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Rebecca Paul, Dr., Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/392-31
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Obesity; Hormone Disturbance; Quality of Life; Hyperandrogenism
Keywords: Bariatric surgery; Sex hormones; Women; Quality of life
MeSH Terms: conditions — Obesity; Endocrine System Diseases; Hyperandrogenism

STUDY DESIGN:
Intervention Model Description: With-in group comparison of pre- and postoperative data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery (Other): Participants will be operated using laparoscopic gastric bypass surgery.
  Interventions: Procedure: Laparoscopic gastric-bypass surgery

INTERVENTIONS:
Procedure: Laparoscopic gastric-bypass surgery — Female participants with BMI >30, between age 18-50, will be operated with laparoscopic gastric bypass surgery by an experienced gastric bypass surgeon.

SUMMARY:
The purpose of this study is to characterize the hormonal status in fertile women undergoing laparoscopic gastric bypass, pre- and postoperatively, and evaluate if there is a correlation between health-related quality of life and proposed hormone changes post-operatively.

DETAILED DESCRIPTION:
Sex hormone levels in women with obesity are altered in comparison to normal weight subjects. Most previous studies have focused on questionnaire surveys, and on the emotional/psychological aspect of health-related quality of life (HRQoL). It has been shown that bariatric surgery can affect reproductive ability, but the relationship between hormonal changes and HRQoL has been sparsely studied.

Hormone balance is affected by fat allocation, insulin levels and liver function, and these factors are all influenced postoperatively. Also body image and altered body mass composition can influence sexuality in diverse ways.

This leads us to theorize that liver production of SHBG will change after surgery and impact serum concentrations of sex hormones. Normalized levels of testosterone and estrogen may lead to reduced symptoms of hyperandrogenism, restitution of normal menstrual cycles and changes in sexual functioning.

The focus of this study is to analyze sexual and health-related quality of life through questionnaire analyses, and to investigate levels of sex hormones pre- and postoperatively in women undergoing bariatric surgery. Results from questionnaire analyses and hormone data will be tested for possible correlations.

ELIGIBILITY:
Inclusion Criteria:

* Premenpausal women
* BMI >30
* Undergoing laparoscopic gastric bypass surgery

Exclusion Criteria:

* Smoking
* Liver disease
* Concomitant hormone treatment including all forms of hormone-based contraception

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biological female.
Enrollment: 68 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Sex-hormone levels | 1 year
  Albumin, luteinizing hormone (LH), follicle stimulating hormone (FSH), sexual hormone binding globulin (SHBG), estradiol (E2), testosterone and progesterone were analyzed preoperatively, and one-year postoperatively.
Female sexual function | 1 year
  A survey of sexual function, the Female Sexual Function Index (FSFI), measures five separate domains of female sexual function: desire/arousal, lubrication, orgasm, satisfaction, and pain. These are assessed as desire (range 1.2-6); arousal (range 0-6); lubrication (range 0-6); orgasm (range 0-6); satisfaction (range 0.8-6) and pain (range 0.6-6). The separate domain scores are summed to create a total score with range 2-36, where totals less than 26 indicate female sexual dysfunction.
Hormone-related quality of life | 1 year
  The Women's Health Questionnaire (WHQ) was developed to assess hormonally-mediated changes that can occur during menopause, but also in other diseases that cause hormonal fluctuation. The following domains are covered by the questionnaire: depressed mood (6 items), somatic symptoms (7 items), anxiety/fears (4 items), vasomotor symptoms (2 items), sleep problems (3 items), sexual behavior (3 items), menstrual symptoms (4 items), memory/concentration (3 items) and attractiveness (3 items). The WHQ is scored by reducing the four point scales (yes definitely, yes sometimes, no not much, no not at all) to binary options (0/1) and the subscale items are summated and divided by the number of items in each subscale. The WHQ questionnaire scores range between zero and one. Zero reflects good health, and one, at the other end of the scale, shows negative health.
Health-related quality of life | 1 year
  The Psychological General Well-Being Survey (PGWB) was developed for the evaluation of perceived well-being and distress and is a 22 item instrument with six domains. Anxiety (range 0-25); Depressed Mood (range 0-15); Positive Well-Being (range 0-20); Self Control (range 0-15); General Health (range 0-15) and Vitality (range 0-20). Scores are summed giving a score range of 22-132, with lower scores indicating poorly perceived well-being.

SECONDARY OUTCOMES:
Correlation between hormone levels and questionnaire results. | 1 year
  Analysis of possible correlations between the change in hormone levels and survey scores 1-year postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Wirén, M.D., PhD., Principal Investigator — Department of Surgery and Department of Clinical and Experimental Medicine, Linköping University, Sweden.

IPD SHARING:
Plan to Share IPD: No
De-indentified individual participant data can be made available for primary and secondary outcomes, upon request, after study completion and manuscript publication.

REFERENCES:
- [Background] Tchernof A, Despres JP. Pathophysiology of human visceral obesity: an update. Physiol Rev. 2013 Jan;93(1):359-404. doi: 10.1152/physrev.00033.2011. PMID 23303913
- [Background] Tchernof A, Despres JP. Sex steroid hormones, sex hormone-binding globulin, and obesity in men and women. Horm Metab Res. 2000 Nov-Dec;32(11-12):526-36. doi: 10.1055/s-2007-978681. PMID 11246820
- [Background] Kolotkin RL, Binks M, Crosby RD, Ostbye T, Gress RE, Adams TD. Obesity and sexual quality of life. Obesity (Silver Spring). 2006 Mar;14(3):472-9. doi: 10.1038/oby.2006.62. PMID 16648619
- [Background] Sarwer DB, Lavery M, Spitzer JC. A review of the relationships between extreme obesity, quality of life, and sexual function. Obes Surg. 2012 Apr;22(4):668-76. doi: 10.1007/s11695-012-0588-1. PMID 22293982
- [Background] Esposito K, Ciotola M, Giugliano F, Bisogni C, Schisano B, Autorino R, Cobellis L, De Sio M, Colacurci N, Giugliano D. Association of body weight with sexual function in women. Int J Impot Res. 2007 Jul-Aug;19(4):353-7. doi: 10.1038/sj.ijir.3901548. Epub 2007 Feb 8. PMID 17287832
- [Background] Gosman GG, King WC, Schrope B, Steffen KJ, Strain GW, Courcoulas AP, Flum DR, Pender JR, Simhan HN. Reproductive health of women electing bariatric surgery. Fertil Steril. 2010 Sep;94(4):1426-1431. doi: 10.1016/j.fertnstert.2009.08.028. Epub 2009 Oct 7. PMID 19815190
- [Background] Malik SM, Traub ML. Defining the role of bariatric surgery in polycystic ovarian syndrome patients. World J Diabetes. 2012 Apr 15;3(4):71-9. doi: 10.4239/wjd.v3.i4.71. PMID 22532886
- [Background] Bond DS, Wing RR, Vithiananthan S, Sax HC, Roye GD, Ryder BA, Pohl D, Giovanni J. Significant resolution of female sexual dysfunction after bariatric surgery. Surg Obes Relat Dis. 2011 Jan-Feb;7(1):1-7. doi: 10.1016/j.soard.2010.05.015. Epub 2010 Jun 4. PMID 20678969
- [Background] Botwood N, Hamilton-Fairley D, Kiddy D, Robinson S, Franks S. Sex hormone-binding globulin and female reproductive function. J Steroid Biochem Mol Biol. 1995 Jun;53(1-6):529-31. doi: 10.1016/0960-0760(95)00108-c. PMID 7626505
- [Background] Sarwer DB, Spitzer JC, Wadden TA, Mitchell JE, Lancaster K, Courcoulas A, Gourash W, Rosen RC, Christian NJ. Changes in sexual functioning and sex hormone levels in women following bariatric surgery. JAMA Surg. 2014 Jan;149(1):26-33. doi: 10.1001/jamasurg.2013.5022. PMID 24190440